CLINICAL TRIAL: NCT01215500
Title: A Study of Dose Escalation of Hypofractionated Radiation Therapy in Patients With Metastatic Cancer
Brief Title: Dose Escalation of Hypofractionated Radiation Therapy in Patients With Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13619B
Record Dates: First submitted 2010-08-02; First posted 2010-10-06 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Tumor; Cancer; Melanoma; Sarcoma; Carcinoma
Keywords: solid tumor cancer; epithelial carcinoma
MeSH Terms: conditions — Neoplasms; Melanoma; Sarcoma; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation therapy (Experimental)
  Interventions: Radiation: Hypofractionated RT

INTERVENTIONS:
Radiation: Hypofractionated RT — RT to site of metastatic disease for three fractions separated by 3 to 8 days. Doses of radiation will increase as follows in order to determine the MTD in Gy:
  For all sites the dose levels are as follows:
  1. 8 Gy/ fraction x 3 fractions = 24 Gy
  2. 10 Gy/fraction x 3 fractions = 30 Gy
  3. 12 Gy/fraction x 3 fractions = 36 Gy
  4. 14 Gy/fraction x 3 fractions = 42 Gy
  5. 16 Gy/fraction x 3 fractions = 48 Gy
  6. 18 Gy/fraction x 3 fractions = 52 Gy
  7. 20 Gy/fraction x 3 fractions = 60 Gy

SUMMARY:
Patients with metastatic cancer are generally treated with chemotherapy, which has improved median survival compared to best supportive care. Despite this, patients continue to have persistent disease at sites that were initially involved with cancer. Radiation therapy is an effective modality for treating localized cancer but generally has been only used for palliation of symptoms once a patient develops metastatic disease. Since patients often have persistent disease after chemotherapy, the goal of this trial is to use increasing doses of radiation therapy to all sites of involved disease in order to determine the safety and efficacy of hypofractionated radiation therapy.

The purpose of this study is to establish a maximum tolerated dose, dose-limiting toxicities, and recommended phase 2 dose of hypofractionated radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of cancer (including epithelial carcinoma, sarcoma, and melanoma)
* Age 18 years and older
* Life expectancy of > 3 months
* Patients with AJCC (6th edition, 2002) stage IV cancer with distant metastases and without pleural or pericardial effusion at diagnosis and before start of study
* Patients with 1-5 sites of maximum tumor dimension (for each individual site) of ≤ 10 cm or < 500 cc volume and amenable to radiation therapy as seen on standard imaging
* Unidimensionally measurable disease (based on RECIST) is desirable but not strictly required
* Brain metastases must have been treated prior to enrollment on study, preferably with stereotactic radiosurgery
* ECOG performance status ≤ 2 or Karnofsky Performance Status ≥ 60%
* No prior radiation therapy to currently involved tumor sites
* Room air saturation > 90%
* Hemoglobin > 9.0 g/dl
* ANC >=1,500/microliter
* Platelets >=100,000/microliter
* Total bilirubin within institutional limits
* Albumin > 2.9 g/dl
* Alkaline phosphatase < 2.5x upper limit of normal
* AST and ALT < 2.5 x upper limit of normal
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Uncontrolled intercurrent illness
* Patients with clinically significant pulmonary dysfunction, cardiomyopathy, or any history of clinically significant CHF are excluded. Exclusion of patients with active coronary heart disease will be at the discretion of the attending physician
* Patients with significant atelectasis such that CT definition of gross tumor volume is difficult to determine
* Pregnancy or breast feeding
* Patients must have no uncontrolled active infection other than that not curable with treatment of their cancer.
* Patients may not be receiving any other investigational drugs during RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-01; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities | 30-90 days
  The dose limiting toxicities occurring within the initial observation period will be defined.
maximum tolerated dose of hypofractionated RT | 30-90 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chmura, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States